CLINICAL TRIAL: NCT03668171
Title: Mesenchymal Stem Cell Transplantation for Acute-on-chronic Liver Failure, a Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Mesenchymal Stem Cell Transplantation for Acute-on-chronic Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Prof. Dr., Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20172049-1
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute-On-Chronic Liver Failure, mesenchymal stem cell,
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be blinded to participant, care provider, investigator and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC group (Experimental): mesenchymal stem cell transplantation via peripheral vein: 0.1-1x10E6 MSCs/kg body weight administered via peripheral vein at week 0, 1, 2 weeks
  Interventions: Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein
- control (Placebo Comparator): placebo infusions (placebo infusion differs from the experimental infusion in only that placebo has no mesenchymal stem cells) will be administered via peripheral vein at week 0, 1, 2
  Interventions: Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein

INTERVENTIONS:
Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein — 0.1-1x10E6 MSCs/kg body weight will be administered via peripheral vein for 3 times at week 0, 4 and 8 mesenchymal stem cell mesenchymal stem cell infusion produced by Cell products of National Engineering Research Center(short for CPNERC), Tianjin, China For control group, placebo infusions will be given to the participants at the same time points

SUMMARY:
Mesenchymal stem cells (MSC) has been reported to improved outcomes of acute-on-chronic liver failure(ACLF). More randomization controlled studies are needed to confirm the effect of MSC treatment for ACLF. This study aimed to investigate the efficacy of mesenchymal stem cells in ACLF patients. This study is an double-blind multicenter randomized and placebo-controlled study. Patients with with ACLF will be randomly assigned to receive MSC treatment (experimental) or standard medical treatment (control). Three times of MSC infusion (0.1-1x10E6cells/kg body weight) via peripheral vein will be given to the experimental group (once per week). The primary outcome is 12 week mortality. Secondary outcomes are clinical remission rate and changes of liver function indices and liver function scores.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years old
* Meeting the criteria of ACLF defined as: 1. definitive chronic liver diseases, acute decompensation within 4 weeks; 2. Significant GI symptom as such fatigue, jaundice,; 3. total bilirubin (TBIL) ≥170 µmo1/L or daily increase of TBIL ≥17.1 µmo1/L; 4. PTA≤40% or INR≥ 1.5; 5. Decompensation of liver functions such as ascites or hepatoencephalopathy;
* MELD score between 17-30. (MELD(i) = 0.957 × ln(Cr) + 0.378 × ln(bilirubin) + 1.120 × ln(INR) + 0.643)
* Chronic liver disease with definitive etiology such as viral hepatitis, alcohol liver disease, drug induced liver injury or autoimmune liver diseases
* Informed consent

Exclusion Criteria:

* Sever complications with 30 days ( GI bleeding, severe infection)；

  --liver cancer or other malignancies
* patients on liver transplantation list
* patients with uncontrolled infections
* severe renal failure
* Severe chronic obstructive pulmonary disease COPD (GOLD III-IV)
* Extrahepatic cholanstasis patients due to biliary obstruction.
* HIV infection
* Pregnant or breast-feeding females.
* Enrolled in other clinical trials with 3 months
* other conditions considered inappropriate for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: 12 week mortality rate | 12 weeks
  mortality rate assessed at week 12

SECONDARY OUTCOMES:
Clinical remission rate at week 12 | 12 weeks
  Clinical remission define as: significant improvement of symptoms and resolution of hepatoencephalopathy; TBIL decrease to below 5 times of ULN，PTA>40% or INR<1.6

CONTACTS AND LOCATIONS:
Locations (1):
- Changcun Guo, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis processes and clinical data of individual participants will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: within 12 months after the study completion and before publications of the findings.